CLINICAL TRIAL: NCT00150345
Title: Immediate vs. Deferred Empirical Antifungal Treatment With Voriconazole In High-Risk Neutropenic Patients With Fever And A Positive Panfungal Polymerase Chain Reaction Assay (IDEA Study)
Brief Title: Immediate vs. Deferred Empirical Antifungal Treatment With Voriconazole In Neutropenic Patients
Acronym: IDEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Infectious Diseases Working Party (AGIHO) of the German Society of Hematology and Oncology (DGHO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1501029
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Possible Fungal Infection
Keywords: Neutropenia; Fever of unknown origin; Empirical treatment; Voriconazole
MeSH Terms: conditions — Neutropenia; Fever of Unknown Origin | interventions — Voriconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early treatment (Experimental): Voriconazole starts within 18 hours of onset of fever intravenously with a loading dose of 6 mg/kg q12h for the first two doses followed by 4 mg/kg q12h (maintenance dose). Switched to oral treatment (200 mg BID) is possible after at least four days. Treatment will be ended if the patient is afebrile (< 38.0 °C) for 7 days with neutrophil counts < 500/µL, or if the patient is afebrile (< 38.0 °C) for 2 days with neutrophil counts > 500/µL.
  Interventions: Drug: voriconazole (Vfend)
- Deferred treatment (Other): Treatment with voriconazole (for dosage see "early treatment arm") is initiated only if a patient is persistently febrile on day 5 after the onset of fever despite antibiotic treatment.
  Interventions: Drug: voriconazole (Vfend)

INTERVENTIONS:
Drug: voriconazole (Vfend) — voriconazole, early treatment
  Arms: Early treatment
Drug: voriconazole (Vfend) — voriconazole, deferred treatment
  Arms: Deferred treatment

SUMMARY:
A well-known side-effect of cytostatics (drugs against malignancies) is a decrease in the number of white blood cells, especially of the so-called neutrophil granulocytes, which are very important for the defense against infections. Hence their decrease (called "neutropenia") leads to a predisposition to infections.

Since infections during neutropenia can be very dangerous, the patients are treated with antibiotics from the very first signs of such an infection (usually fever). If the antibiotics (drugs against bacteria) do not lead to a normalization of the body temperature within four days, a drug against fungi is added.

In the IDEA study, one half of the patients receive the antifungal drug voriconazole (as usual) only in case the antibiotics alone do not lead to a normalization of the body temperature (current standard of care). The other half of the patients receive voriconazole immediately after onset of fever (concomitantly with the antibiotics).

The research question is, whether in the "early-treatment" group fewer manifest fungal infections will be observed than in the "late-treatment" group.

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia, aggressive lymphoma, bone marrow or stem cell transplantation;
* Neutropenia (<500 neutrophils/µL) of at least 10 days;
* Newly diagnosed fever;
* Positive panfungal polymerase chain reaction assay

Exclusion Criteria:

* Documented bacterial infection during screening or at randomization
* Fungemia or other documented invasive fungal infection during screening or at randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2005-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- Germany (25):
  - Pfizer Investigational Site, Augsburg
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bielefeld
  - Pfizer Investigational Site, Bremen
  - Pfizer Investigational Site, Chemnitz
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Frankfurt (Oder)
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Homburg/Saar
  - Pfizer Investigational Site, Kiel
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Ludwigshafen
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Potsdam
  - Pfizer Investigational Site, Stuttgart
  - Pfizer Investigational Site, Trier
  - Pfizer Investigational Site, Wiesbaden
  - Pfizer Investigational Site, Würzburg

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501029&StudyName=Immediate%20vs.%20Deferred%20Empirical%20Antifungal%20Treatment%20With%20Voriconazole%20In%20Neutropenic%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 810 participants screened; 81 assigned to immediate voriconazole treatment and 66 to deferred voriconazole treatment. Study should be considered a pilot study; planned sample size (n=200) was not based on statistical power considerations.
Pre-assignment Details: Screening phase started with cytoreductive treatment; screening phase ended at onset of fever or if reconstitution of leukocytes to >1000 per microliter (1000/uL) or neutrophils to >500/uL. Randomization occurred within 18 hours after onset of fever (if febrile or had positive polymerase chain reaction (PCR) assay prior to onset of fever).
Groups:
- Immediate Voriconazole: Voriconazole intravenous (IV) loading dose of 6 milligrams per kilogram (mg/kg) every 12 hours on Day 1 for the first 2 doses followed by 4 mg/kg IV every 12 hours (maintenance dose) for at least 4 days (up to Day 5). Continued treatment with oral (PO) voriconazole 200 mg twice a day (BID) through Day 28. Treatment ended if the participant was afebrile (< 38.0 degrees Celsius [C]) for 7 days with neutrophil counts < 500 per microliter (500/uL) or if participant was afebrile (< 38.0 degrees C) for 2 days with neutrophil counts > 500/uL.
- Deferred Voriconazole Treatment: Placebo IV loading dose of 6 mg/kg every 12 hours on Day 1 for the first 2 doses followed by 4 mg/kg IV every 12 hours (maintenance dose) for at least 4 days (up to Day 5). On Day 5, voriconazole IV loading dose of 6 mg/kg every 12 hours for at least 4 days (up to Day 9). Continued treatment with PO voriconazole 200 mg BID through Day 28. Treatment ended if the participant was afebrile (< 38.0 degrees C) for 7 days with neutrophil counts < 500/uL or if participant was afebrile (< 38.0 degrees C) for 2 days with neutrophil counts > 500/uL.
Period: Overall Study
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Started | 81 | 66
Completed | 47 | 34
Not Completed | 34 | 32
Not completed — Death | 5 | 2
Not completed — Adverse Event | 8 | 6
Not completed — Lack of Efficacy | 5 | 4
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Laboratory abnormality | 1 | 2
Not completed — Other | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment | Total
Number analyzed (Participants) | 81 | 66 | 147
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 29 | 17 | 46
  Between 45 and 64 years | 31 | 35 | 66
  >=65 years | 21 | 14 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 29 | 68
  Male | 42 | 37 | 79
Race/Ethnicity, Customized [Number; unit: participants]
  White | 81 | 65 | 146
  Other | 0 | 1 | 1
Weight [Mean (Full Range); unit: kilograms (kg)] | 77.1 [42.0 to 112.5] | 79.2 [45.3 to 152.0] | 78.1 [42.0 to 152.0]
Height [Mean (Full Range); unit: centimeters (cm)] | 172.1 [150.0 to 196.0] | 171.9 [153.0 to 198.0] | 172.0 [150.0 to 198.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Proven or Probable Invasive Fungal Infections (IFI): Complete Case Analysis
Description: Number of participants with proven (deep tissue infection, fungemia, or endemic fungal infections) or probable IFI (at least 1 host criterion [fever, body temperature <36 or >38 degrees Celsius, graft-versus-host disease, use of corticosteroids]; and 1 microbiological criterion [fungal or yeasts]; or clinical criteria [abnormal site consistent with infection]) as defined by European Organization for Research and Treatment of Cancer Mycosis Study Group (EORTC/MSG) criteria. Complete case analysis: must be evaluable until Day 28 or had developed a proven or probable IFI by the final visit.
Time Frame: Day 2 through Day 28
Population: Modified Intent-to-Treat population (MITT): participants in ITT population (at least 1 dose of study treatment) with valid post-baseline proven or probable IFI, did not have fungemia or other IFI at screening or randomization, no antipyretic analgesics on Day 5 (or Day 9 of open-label voriconazole). N=number of complete case evaluable participants.
Measure: Number; unit: participants
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 43 | 35
participants | 6 | 9
Statistical Analysis 1: Comparison: Immediate Voriconazole vs Deferred Voriconazole Treatment; Hypothesis: H0: rv - rp = 0 vs H1: rv - rp does not equal 0, where ri is rate of IFI (i=v for voriconazole group, i=p for deferred voriconazole group). Logit model (including important covariates) used. The adjusted odds ratio and 95 percent (%) confidence interval (CI) for adjusted odds ratio calculated. If 95% CI around odds ratio does not contain a value of 1, then the null hypothesis of equal rates of IFI between immediate voriconazole and deferred voriconazole to be rejected; Test type: Superiority or Other; p = 0.258, Regression, Logistic; Odds Ratio (OR) = 0.493, 95% CI 2-sided [0.129 to 1.755] — Odds ratio computed from the logistic regression (logit model) including terms for treatment arm, concomitant fluconazole, and positive PCR before randomization. Event IFI=yes is modeled

2. Secondary Outcome: Number of Participants With Defervescence Day 5 (4 Days After Initiation of Study Treatment)
Description: Number of participants who achieved defervescence (were afebrile). Defervescence stated if all of a participants's body temperatures within 24 hours of evaluation time were <38.0 degrees C. Defervescence was not stated and participant was discontinued from the study if participant received antipyretics (non-steroidal anti-inflammatory drugs or paracetamol).
Time Frame: Day 5 (96 hours through 120 hours after start of study treatment)
Population: MITT
Measure: Number; unit: participants
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
participants | 32 | 28
Statistical Analysis 1: Comparison: Immediate Voriconazole vs Deferred Voriconazole Treatment; Test type: Superiority or Other; p = 0.596, Regression, Logistic; Odds Ratio (OR) = 0.822, 95% CI 2-sided [0.398 to 1.696] — Odds ratio computed from the logistic regression (logit model) including terms for treatment arm, concomitant fluconazole, and positive PCR before randomization. Event defervescence=yes is modeled

3. Secondary Outcome: Number of Participants With Defervescence Day 9 (8 Days After Initiation of Study Treatment)
Description: Number of participants who achieved defervescence (were afebrile). Defervescence stated if all of a participant's body temperatures within 24 hours of evaluation time were <38.0 degrees C. Defervescence was not stated and participant was discontinued from the study if participant received antipyretics (non-steroidal anti-inflammatory drugs or paracetamol).
Time Frame: Day 9 (192 hours through 216 hours after start of study treatment)
Population: MITT
Measure: Number; unit: particpants
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
particpants | 42 | 34
Statistical Analysis 1: Comparison: Immediate Voriconazole vs Deferred Voriconazole Treatment; Test type: Superiority or Other; p = 0.864, Regression, Logistic; Odds Ratio (OR) = 0.936, 95% CI 2-sided [0.441 to 1.988] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Time to Continuous Defervescence
Description: Time (in days) from start of study medication to continuous defervescence. Continuous defervescence stated if participant maintains a body temperature of <38.0 degrees C for at least 96 hours.
Time Frame: Day 2 through Day 28
Population: MITT
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
days | 6.0 [4.0 to 8.0] | 5.0 [4.0 to 7.0]
Statistical Analysis 1: Comparison: Immediate Voriconazole vs Deferred Voriconazole Treatment; Test type: Superiority or Other; p = 0.955, Log Rank

5. Secondary Outcome: Number of Participants Per Reason for Lack of Defervescence
Time Frame: Day 2 through Day 28
Population: MITT
Measure: Number; unit: participants
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
participants
  Fungal infection | 3 | 3
  Bacterial infection | 7 | 6
  Viral infection | 1 | 0
  Unknown | 4 | 4
  Other | 3 | 3
  Missing evaluation response | 0 | 1

6. Secondary Outcome: Number of Participants That Died on or Before Day 28 (Mortality)
Description: Number of participants that died on or before Day 28 after start of study treatment. A participant must be evaluable until Day 28 (final visit) or have died before the final visit.
Time Frame: Day 2 through Day 28
Population: MITT; N=number of participants evaluable until Day 28 (final visit) or died before the final visit.
Measure: Number; unit: participants
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 43 | 29
participants | 4 | 1
Statistical Analysis 1: Comparison: Immediate Voriconazole vs Deferred Voriconazole Treatment; Difference in proportions expressed as a percent: immediate voriconazole versus (vs) deferred voriconazole treatment; Test type: Superiority or Other; Difference in % participants that died = 5.85, 95% CI 2-sided [-5.08 to 16.78] — Approximate 2-sided confidence interval (CI)

7. Secondary Outcome: Time to Negative Panfungal Polymerase Chain Reaction (PCR)
Description: Time (in days) from start of study medication to negative panfungal PCR; assessed for participants whose most recent panfungal PCR result prior to start of study medication was positive. Defined as negative if at least 2 successive and all following panfungal PCR assessments from start of study medication until 24 hours after end of treatment are negative. Measured as first quartile of time (point in time measurement; no median or measure of dispersion calculated); median time was not estimable for deferred voriconazole treatment group.
Time Frame: Day 2 through Day 28
Population: MITT; N=number of participants whose most recent panfungal PCR result prior to start of study medication was positive.
Measure: Number; unit: days
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 10 | 8
days | 4.0 | 5.5
Statistical Analysis 1: Comparison: Immediate Voriconazole vs Deferred Voriconazole Treatment; Test type: Superiority or Other; p = 0.190, Log Rank

8. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association of Positive PCR Assessments With Achievement of Continuous Defervescence (Yes)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with achievement of continuous defervescence (response=Yes). Continuous defervescence stated if participant maintains a body temperature of <38.0 degrees C for at least 96 hours. Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: MITT; N=number of participants who completed the study and had a non-missing value for percent of positive panfungal PCR.
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 36 | 27
percent of positive PCR assessments | 10.6 (14.11) | 8.0 (14.71)
Statistical Analysis 1: Comparison: Immediate Voriconazole vs Deferred Voriconazole Treatment; Continuous defervescence achieved=Yes; Test type: Superiority or Other; p = 0.049, Regression, Linear — SAS PROC REG with SELECTION=STEPWISE option of SLENTRY=0.05 and SLSTAY=0.10 utilized. Stepwise option combined forward stepping (with a 0.05 level to enter) with elimination of variables already in model that do not stay significant at 0.10 level; Variables: association with age, c-reactive protein, and time to continuous defervescence not significant at 0.05 level; not included in final model; Mean Difference (Final Values) = -22.031, 95% CI 2-sided [-44.004 to -0.059], Standard Error of Mean 10.888

9. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association of Positive PCR Assessments With Achievement of Continuous Defervescence (No)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with achievement of continuous defervescence (response=No). Continuous defervescence stated if participant maintains a body temperature of <38.0 degrees C for at least 96 hours. Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 3 | 0
percent of positive PCR assessments | 21.7 (20.21) |

10. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Age
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with age for participants who completed the study and have a non-missing value for percent of positive panfungal PCR.
Time Frame: Day 2 through Day 28
Population: MITT. Correlation of positive panfungal PCR assessments with age was not summarized as planned.
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Gender
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with gender (Female or Male). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: MITT; (n)=number of participants who completed the study and had a non-missing value for percent of positive panfungal PCR for immediate voriconazole and deferred voriconazole treatment, respectively.
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Female (n=21, 12) | 12.3 (14.82) | 4.2 (10.36)
  Male (n=18, 15) | 10.4 (14.75) | 11.1 (17.16)

12. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Primary Underlying Neoplastic Disease
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with primary underlying neoplastic disease. Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Acute lymphatic leukemia (n=6, 6) | 13.9 (16.39) | 9.7 (15.29)
  Acute myeloid leukemia (n=29, 18) | 10.5 (14.39) | 8.8 (15.78)

13. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Planned Allogeneic Transplants
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with allogeneic bone marrow transplant or allogeneic peripheral stem cell transplant (Yes or No). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Association Yes (n=13, 9) | 10.5 (14.88) | 6.5 (13.03)
  Association No (n=26, 18) | 11.9 (14.77) | 8.8 (15.78)

14. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Concomitant Fluconazole
Description: Percent positive panfungal PCR assessments during treatment phase of study in association with use of concomitant (prophylaxis) fluconazole (Yes or No). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Association Yes (n=8, 4) | 13.5 (15.39) | 6.3 (12.50)
  Association No (n=31, 23) | 10.9 (14.63) | 8.3 (15.28)

15. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Neutrophil Count >500 uL
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with neutrophil count >500 uL (Yes or No). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Association Yes (n=24, 20) | 10.9 (14.60) | 7.9 (15.17)
  Association No (n=15, 7) | 12.3 (15.13) | 8.3 (14.43)

16. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With C-reactive Protein Level >1.25 Times the Upper Limit of Normal (x ULN)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with c-reactive protein level (measured in milligrams per liter [mg/L]) >1.25 x ULN (Yes or No). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: MITT. Correlation of positive panfungal PCR assessments with c-reactive protein level was not summarized as planned.
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Fungal Species Identified
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with fungal species (singular [one species]=sp; plural [many species]=spp) identified (Yes or No). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Aspergillus flavus: No (n=39, 27) | 11.4 (14.62) | 8.0 (14.71)
  Aspergillus fumig: No (n=38, 27) | 11.7 (14.70) | 8.0 (14.71)
  Aspergillus nidulans: No (n=39, 27) | 11.4 (14.62) | 8.0 (14.71)
  Aspergillus sp: No (n=39, 27) | 11.4 (14.62) | 8.0 (14.71)
  Aspergillus spp: No (n=37, 27) | 11.6 (14.88) | 8.0 (14.71)
  Candida albicans: Yes (n=2, 4) | 16.7 (23.57) | 0.0 (0.0)
  Candida albicans: No (n=37, 23) | 11.2 (14.45) | 9.4 (15.55)
  Candida glabrata: Yes (n=2, 1) | 33.3 (0.00) | 0.0 (0.0)
  Candida glabrata: No (n=37, 26) | 10.3 (14.06) | 8.3 (14.91)
  Candida krusei: No (n=39, 26) | 11.4 (14.62) | 8.3 (14.91)
  Candida spp: No (n=38, 27) | 11.7 (14.70) | 8.0 (14.71)
  Candida tropicalis: No (n=39, 27) | 11.4 (14.62) | 8.0 (14.71)

18. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Fungal Species Identified (Aspergillus Spp=Yes)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with fungal species (singular [one species]=sp; plural [many species]=spp) identified (Yes). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 2 | 0
percent of positive PCR assessments | 8.3 (11.79) |

19. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Proven or Probable IFI (Complete Cases) Between Day 2 and Day 28
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with proven or probable IFI (complete cases) between Day 2 and Day 28 (Yes or No). Complete case analysis: participant must be evaluable until Day 28 (final visit) or have developed a proven or probable IFI by the final visit. Participant considered evaluable until Day 28 if participant completed the study and completed an assessment of IFI at Day 28 or final visit. Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Association Yes (n=2, 2) | 0.0 (0.0) | 16.7 (23.57)
  Association No (n=37, 25) | 12.1 (14.77) | 7.3 (14.30)

20. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Defervescence Day 5 (4 Days After Initiation of Study Treatment)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with defervescence (were afebrile) Day 5 (Yes or No). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 5 (96 hours through 120 hours after start of study treatment)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Groups:
- Deferred Voricoazole Treatment: Placebo IV loading dose of 6 mg/kg every 12 hours on Day 1 for the first 2 doses followed by 4 mg/kg IV every 12 hours (maintenance dose) for at least 4 days (up to Day 5). On Day 5, voriconazole IV loading dose of 6 mg/kg every 12 hours for at least 4 days (up to Day 9). Continued treatment with PO voriconazole 200 mg BID through Day 28. Treatment ended if the participant was afebrile (< 38.0 degrees C) for 7 days with neutrophil counts < 500/uL or if participant was afebrile (< 38.0 degrees C) for 2 days with neutrophil counts > 500/uL.
Arm/Group | Immediate Voriconazole | Deferred Voricoazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Association Yes (n=28, 21) | 14.5 (14.58) | 8.3 (15.81)
  Association No (n=11, 6) | 3.6 (12.06) | 6.9 (11.08)

21. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Defervescence (Yes) by Day 9 (8 Days After Initiation of Study Treatment)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with defervescence (were afebrile) Day 9 (Yes). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 9 (192 hours through 216 hours after start of study treatment)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 37 | 27
percent of positive PCR assessments | 11.0 (14.11) | 8.0 (14.71)

22. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Defervescence (No) by Day 9 (8 Days After Initiation of Study Treatment)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with defervescence (were afebrile) Day 9 (No). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 9 (192 hours through 216 hours after start of study treatment)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 2 | 0
percent of positive PCR assessments | 20.0 (28.28) |

23. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Time to Defervescence
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with time to defervescence. Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: MITT. Correlation of positive panfungal PCR assessments with time to defervescence was not summarized as planned.
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Reasons for Lack of Continuous Defervescence (No)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with lack of continuous defervescence (No). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
percent of positive PCR assessments
  Fungal infection: No (n=39, 27) | 11.4 (14.62) | 8.0 (14.71)
  Bacterial infection: No (n=39, 27) | 11.4 (14.62) | 8.0 (14.71)
  Viral infection: No (n=39, 27) | 11.4 (14.62) | 8.0 (14.71)
  Unknown infection: No (n=36, 27) | 10.6 (14.11) | 8.0 (14.71)
  Other infection: No (n=39, 27) | 11.4 (14.62) | 8.0 (14.71)

25. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Reasons for Lack of Continuous Defervescence: Unknown Infection (Yes)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with lack of continuous defervescence (Yes). Percent calculated as number of positive PCR assessments divided by number of all PCR assessments in treatment phase multiplied by 100.
Time Frame: Day 2 through Day 28
Population: MITT; N=number of participants who completed the study and had a non-missing value for percent of positive panfungal PCR for immediate voriconazole and deferred voriconazole treatment, respectively.
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 3 | 0
percent of positive PCR assessments | 21.7 (20.21) |

26. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Mortality by Day 28 (Alive)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with mortality on or before Day 28 after start of study treatment (Alive). A participant must be evaluable until Day 28 (final visit).
Time Frame: Day 2 through Day 28
Population: MITT; participants who completed the study and had a non-missing value for percent of positive panfungal PCR. N=number of participants for category "Alive".
Measure: Mean (Standard Deviation); unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 39 | 27
percent of positive PCR assessments | 11.4 (14.62) | 8.0 (14.71)

27. Secondary Outcome: Course of Positive Panfungal PCR Assessments to Explanatory Variables: Association With Mortality by Day 28 (Died)
Description: Percent of positive panfungal PCR assessments during treatment phase of study in association with mortality on or before Day 28 after start of study treatment (Died). A participant must have died before Day 28 (final visit).
Time Frame: Day 2 through Day 28
Population: MITT; participants who completed the study and had a non-missing value for percent of positive panfungal PCR: no participants met this criteria within the category "Died".
Measure: Number; unit: percent of positive PCR assessments
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Number of Participants Assessed as Needing Further Antineoplastic Therapy as Planned
Time Frame: Day 28
Population: MITT
Measure: Number; unit: participants
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 68 | 54
participants | 42 | 32
Statistical Analysis 1: Comparison: Immediate Voriconazole vs Deferred Voriconazole Treatment; Difference in proportions expressed as a percent: immediate voriconazole vs deferred voriconazole treatment; Test type: Superiority or Other; Difference in percentages = 2.51, 95% CI 2-sided [-14.96 to 19.97]

29. Secondary Outcome: Number of Participants With Reasons Why Antineoplastic Therapy Not Continued as Planned
Time Frame: Day 28
Population: MITT; data not summarized as planned; data insufficient for analysis due to missing data.
Measure: Number; unit: participants
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 7 days after last dose of study drug
Description: Safety population = all randomized participants with at least 1 dose of study treatment. The same event may appear as both an AE and SAE; however, they are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Immediate Voriconazole | Deferred Voriconazole Treatment
Serious Adverse Events (participants affected / at risk) | 8/81 | 8/66
Other Adverse Events (participants affected / at risk) | 58/81 | 38/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Voriconazole (N=81) | Deferred Voriconazole Treatment (N=66)
Coronary artery disease (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Encephalitic infection (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Mucormycosis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Voriconazole (N=81) | Deferred Voriconazole Treatment (N=66)
Visual impairment (Eye disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 7 | 3
Diarrhoea (Gastrointestinal disorders) | 22 | 13
Nausea (Gastrointestinal disorders) | 12 | 6
Vomiting (Gastrointestinal disorders) | 9 | 5
Chest pain (General disorders) | 2 | 5
Mucosal inflammation (General disorders) | 7 | 3
Oedema (General disorders) | 5 | 3
Oedema peripheral (General disorders) | 6 | 1
Pyrexia (General disorders) | 7 | 5
C-reactive protein increased (Investigations) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 2
Headache (Nervous system disorders) | 8 | 11
Hallucination (Psychiatric disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Rash (Skin and subcutaneous tissue disorders) | 14 | 6
Hypertension (Vascular disorders) | 5 | 3

LIMITATIONS AND CAVEATS:
One participant in the Immediate Voriconazole treatment group was incorrectly included in the original Primary efficacy analysis and has now been excluded; IFI was identified on the day study treatment started (not prior to study treatment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.